CLINICAL TRIAL: NCT00629395
Title: Computerized Cognitive Training for Childhood Cancer Survivors: A Pilot Study
Brief Title: Computerized Cognitive Training for Childhood Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00001502
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Primary Brain Tumor
Keywords: pediatric; brain tumor; survivors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Participate in 12 week computer program.
  Interventions: Behavioral: Captain's Log Computer Program

INTERVENTIONS:
Behavioral: Captain's Log Computer Program — 12 Computer Program

SUMMARY:
Specific Aim 1: To assess the feasibility and acceptability of a home-based, computerized attention training program with survivors of central nervous system (CNS) impacting pediatric cancer (e.g. acute lymphocyte leukemia [ALL], brain tumors).

Specific Aim 2: To estimate the effect size of this attention training program with survivors of childhood cancer to determine whether a larger-scale clinical trial is warranted.

DETAILED DESCRIPTION:
Pediatric patients meeting initial eligibility criteria will be identified through the databases for each clinic (n = approximately 50 survivors in each clinic). A letter explaining the purpose of the study will then be sent to the parents of these patients. Interested parents will be invited to contact study personnel by phone or email for a thorough review of the study and to schedule a screening appointment.

After obtaining written informed consent and assent (from parents and child, respectively), screening procedures will include administration of an abbreviated intellectual test battery, two working memory tasks, and a computerized attention measure to the survivor. Parents will complete questionnaire measures regarding their child's adaptive, behavioral, emotional, and attentional functioning; follow-up interviewing will be conducted to clarify any potential problems identified on the questionnaires. The entire screening procedure is estimated to take approximately 60 minutes for the survivor and 30-45 minutes for parents. To maximize efficiency, a research assistant will complete testing with the child and a psychologist will explain the questionnaire measures to the parent and conduct any follow-up interviewing.

ELIGIBILITY:
Inclusion Criteria:

1. A T-score greater than the 75th percentile on either the Cognitive Problems/Inattention or the DSM-IV Inattention subscales of the Conners' Parent Rating Scale
2. One or more standard deviations below the mean on the Working Memory Index of the WISC-IV or a Working Memory Index that is one or more standard deviations below the participant's estimated IQ.

These criteria are based on the eligibility criteria used in the largest trial to date of psychostimulant methylphenidate (MPH; commonly known as Ritalin) with survivors of childhood cancer.

Exclusion Criteria:

1. Estimated IQ ≤ 70
2. Motor, visual, or auditory handicap that prevents computer use
3. A diagnosis of attention-deficit hyperactivity disorder (ADHD), oppositional defiant disorder (ODD), depression, autism, or pervasive developmental disorder (PDD)
4. Insufficient fluency in English.

Participants who are currently taking stimulant medications (stable dose for at least 30 days) for attentional difficulties, but who meet inclusion criteria will be allowed to participate.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Computer program results | baseline and study completion

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Hardy, PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States